CLINICAL TRIAL: NCT00145834
Title: A Randomised Community Based Experimental Trial in the Health Visitor's Practice Field
Brief Title: Early Breastfeeding Cessation - is It Possible to Prevent?
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Lundbeck Foundation (Other); Sygekassernes Helsefond (Other); Ringkjobing Amt (Unknown); Ribe Amt (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUN-2002-653
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: Breastfeeding; Practice; Maternal Behaviour; Self-Efficacy
Keywords: psychosocial factors; breastfeeding; postnatal intervention; health visitor
MeSH Terms: conditions — Breast Feeding

INTERVENTIONS:
Behavioral: community based trial

SUMMARY:
The purpose of this study is to investigate if a postnatal public health breastfeeding intervention relying on the importance of the psychosocial factors can prolong the period with exclusive breastfeeding duration among mothers who want to breastfeed.

DETAILED DESCRIPTION:
Breastfeeding is a complex learned behaviour and not a capability which comes naturally with motherhood. Different types of professional recommendations have been used to support the new mother in this process.

Randomised studies have shown that postnatal support can influence the breastfeeding duration positively. Various studies has offered different kinds of interventions with home visits and/or telephone calls as the generally used approach, but the proper follow-up on the breastfeeding support in the postnatal period after the mother leaves the hospital is not yet clear.

ELIGIBILITY:
Inclusion Criteria:

* Danish mother, single child, gestational age of not less than 37 full weeks

Exclusion Criteria:

* Mothers with an ethic background other than Danish, preterm delivery,twin birth

Min Age: 0 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 1456
Dates: Start 2004-02; Study Completion 2005-04

PRIMARY OUTCOMES:
Breastfeeding duration

SECONDARY OUTCOMES:
Satisfaction with the breastfeeding period

CONTACTS AND LOCATIONS:
Overall Officials: Ingegerd Harder, Ph.D., Study Director — Department of Nursing Science, University of Aarhus
Locations (1):
- Institute of Publich Health, Department of Nursing Science, University of Aarhus, Aarhus, Denmark